CLINICAL TRIAL: NCT00781755
Title: Phase 4 Study of Treating Schizophrenic Smokers Using Varenicline and Behavioral Intervention: Effects on Craving, Cues and Withdrawal
Brief Title: Treating Schizophrenic Smokers: Effects on Craving, Cues and Withdrawal
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study design was altered such that a treatment component was removed through the VA IRB. We did not and will not begin this clinical trial.
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Gary B. Kaplan, M.D./ Director, Mental Health Service/ Professor of Psychiatry and Pharmacology, VA Boston Healthcare System/ Boston University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1988; VABHS IRB Protocol #1988
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2008-12

CONDITIONS: Tobacco Use Disorder
Keywords: smoking cessation; varenicline; schizophrenia; serious mental illness; Nicotine addiction; Smoking Behavior
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Schizophrenia; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): VAR-MI: This group will receive 1mg/day varenicline (titrated from .5mg/day) and two sessions of a motivational interviewing platform CBT treatment over the course of two weeks.
  Interventions: Drug: varenicline; Behavioral: Adaptation of Motivational Interviewing
- 2 (Placebo Comparator): PLA-MI: VAR-MI: This group will receive a daily placebo pill and two sessions of a motivational interviewing platform CBT treatment over the course of two weeks.
  Interventions: Behavioral: Adaptation of Motivational Interviewing

INTERVENTIONS:
Drug: varenicline — .5mg/day for 3 days then titrated to 1.0mg/day for 11 days. A total dosing regimen of 14 days.
  Arms: 1
Behavioral: Adaptation of Motivational Interviewing — 2 sessions of behavioral intervention designed to create ambivalence about quitting or plan for a quit attempt if the patient is ready.

SUMMARY:
This is a clinical research protocol to study the efficacy of combined varenicline (Chantix) and motivational interviewing (MI) for smoking cessation in a sample of smokers who have been diagnosed with schizophrenia or schizoaffective disorder. The study is a double-blind, randomized, controlled, subacute treatment trial of MI plus varenicline (VAR-MI) versus MI plus placebo (PLA-MI). The pharmaceutical treatment will utilize Chantix at a dose of 1 mg/day for a period of two weeks.

The primary goal is to determine if VAR-MI decreases baseline behavioral measures of urge and withdrawal and reduces baseline rates of cigarette consumption. The primary efficacy measures of VAR-MI vs. PLA-MI treatment are: Minnesota Nicotine Withdrawal Scale, Questionnaire for Smoking Urge-brief, number of cigarettes smoked per day in the previous week, CO levels, and Brief Psychiatric Rating Scale and Positive And Negative Symptom Scale scores on the last day of the study. Other primary outcome measures are to determine the effects of VAR-MI and PLA-MI on smoking cue-induced urges in tobacco cue reactivity sessions and reward responsiveness as assessed by a computerized task.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants for this study:

* Are between the ages 18-65 years of age
* Are daily cigarette smokers
* Have smoked a minimum of 10 cigarettes per day for at least one year
* Are confirmed smokers as verified by CO
* Have a psychiatric diagnosis of schizophrenia or schizoaffective disorder (any subtype) as determined by the SCID-IV. Participants must have received a stable dose of antipsychotic medication for at least 2 weeks prior to beginning the study. Patients receiving clozapine at 500 mg/day or more must also be receiving anti-seizure prophylaxis. Patients must be determined to be psychiatrically stable at baseline as established by standardized interview and medical review by psychiatrist.

Exclusion Criteria:

Individuals who are not eligible to participate in this study include individuals with:

* Any serious or unstable medical problem in the last 6 months
* Severe renal impairment
* A history of clinically significant allergic reactions to nicotine agonist medications
* Current primary use of tobacco products other than cigarettes
* Breath alcohol level > 0.005 g/l at screening
* Current substance abuse or dependence (besides nicotine)
* Current attempts to quit smoking using any method
* Designation as legally incompetent to sign the informed consent (i.e., have a guardian or have delegated power of attorney to another).

Other exclusions are:

* Current use of medications that might affect the behavioral response to cigarette smoking, including transdermal nicotine or nicotine gum and bupropion - Inability to participate in the screening session due to severe psychosis, severe depression or suicidality, current mania, or an organic mental disorder such as dementia or delirium
* Presence of unstable psychiatric symptoms or clinical deterioration (i.e., unstable psychosis, homicidality, or suicidality) within the last month.
* Females of childbearing potential are eligible if not pregnant or nursing and if they practice effective contraception (oral, injectable, or implantable contraceptives; intrauterine device; or barrier method with spermicide).
* There currently are no known contraindications to the use of varenicline and no identified drug-drug interactions. However, reduced dosage of varenicline is recommended for individuals with severe renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Reported Smoking Urge and Withdrawal | 2 weeks

SECONDARY OUTCOMES:
Smoking Status | 2 weeks
Mood Ratings | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary B Kaplan, M.D., Principal Investigator — VA Boston Healthcare System; Suzy Bird Gulliver, Ph.D., Study Chair — VISN 17 Center of Excellence for Research on Returning War Veterans; Barbara W Kamholz, Ph.D., Study Chair — VA Boston Healthcare System; James Levitt, M.D., Study Chair — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System Brockton Medical Center, Brockton, Massachusetts, United States